CLINICAL TRIAL: NCT01640509
Title: A Phase I-II Synchrotron Radiation Application to the Treatment of Intracranial Tumors
Brief Title: Synchrotron Radiation to the Treatment of Intracranial Tumors
Acronym: ESRF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 08 06
Record Dates: First submitted 2012-06-28; First posted 2012-07-13 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Brain Cancer
Keywords: Radiotherapy, Targeted
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- synchrotron radiation (Experimental): treated by synchrotron radiation
  Interventions: Radiation: treated by synchrotron radiation

INTERVENTIONS:
Radiation: treated by synchrotron radiation — treated by synchrotron radiation

SUMMARY:
The purpose of this study is to prove the safety and acceptability of treatment with the Synchrotron radiation by medium-term medical follow-up of the patients.

DETAILED DESCRIPTION:
Synchrotron radiation (SR) is used to produce monochromatic X-ray photons of very high intensity with tunable energy in the range of medium energies (0-150 keV). Thus freed of low energies, the penetration is still important and the types of possible interactions are, in addition to the Compton Effect in water, the photoelectric effect with any atom much heavier than those of the living mater represented by the carbon, oxygen, hydrogen, nitrogen and phosphorus. Photoelectric interactions cause energy deposits much larger than the Compton Effect, but they require the presence of foreign atoms in living tissue to occur. It may be, for example iodine, platinum or gadolinium, all these atoms are commonly introduced into the human body in medical practice as contrast media in radiology, or as anti-neoplastic chemotherapy.

The use of SR for radiotherapy, if you want to take advantage of its original properties, needs the use of a combined treatment: radiation plus medication bringing the heavy atoms suitable for photo electric effect. Such a concept of combined therapy is widely used in radiotherapy for decades and was the source of many advances in treatment, some are presently routine practices (chemo-radiotherapy, photodynamic therapy) other are still under study as translational research (boron neutron capture therapy). The SR photons at these "photoelectric" energy band can cause highly cytotoxic damages in tumors especially when treated with platinum (cisplatin or carboplatin). Indeed, they provide a photoelectric activation of platinum atoms leading to a massive energy deposition in the DNA of tumors. This therapeutic principle has been called platinum photoactivation therapy (PAT-plat). It is particularly suitable for tumors of small to medium volumes, localized small to medium-depth and suitable for a multi-beam ballistics. Also if there is a possibility of loading the tumor tissue with high doses of heavy compounds to achieve the combined treatment in favorable conditions, one would expect a greater therapeutic effect than conventional treatments. Brain tumors represent a model with these features, thanks to recent techniques of convection enhanced delivery (CED), which allow a direct infusion of medication in the tumor.

This work is not conceptually particularly complex although technically sensitive and very original since ESRF and the Grenoble University Hospital are the only institution which have made the effort to date to develop in close cooperation a SR line entirely devoted to biomedical research. There is no other site in the world is this situation, most of the other centers have either lower energies, or do not have the immediate vicinity of an academic medical center that can set up the collaboration needed or are too new to have already reached this experimental level. On the other hand, the technical and material investments are rather important and as information flow is very free, it was not considered appropriate at this time to start such research simultaneously in several sites. The ESRF and the RSRM team ("Rayonnement Synchrotron et Recherche Médicale") are therefore pioneers in this field and their work is well known worldwide. The 2010 Equipex call for tender agreed to fund the first table top synchrotron prototype to be designed and assembled in Orsay : ThomX project at the LAL, laboratoire de l'accélérateur linéaire, our team is associated to this development. Our technique might spread outside the domain of the great instruments [http://sera.lal.in2p3.fr/thomx/]..

To carry out the treatment with a satisfactory distribution of the dose of SR, it is necessary to increase the stopping power of the target tumor by the use of an injection of iodinated contrast medium at the time of irradiation. This treatment can be applied to any tumor having good contrast uptake at CTscan and incidentally which may be treated with platinum. For these reasons, the anatomical location of intracranial human tumors has been chosen for the study of the application of this treatment with SR monochromatic 80 keV.

The experimental treatment will be a part of standard treatment for brain metastases under conformal radiotherapy or stereotactic. This irradiation will complement a pan-encephalic standard irradiation that will be made later, thus providing additional security in terms of dosimetry.

Main objective: To prove the safety and acceptability of treatment with the SR by medium-term medical follow-up of the patients.

Primary outcome: limiting adverse events will be judged according to international scales appropriate to the post-irradiation "acute" toxicity: radiation therapy and / or chemo-radiotherapy NCI-CTC scale; post- irradiation "late" toxicity radiation therapy and / or chemo-radiotherapy SOMA-LENT scale. The acceptable limit for these two criteria will be grade <3; performance status (WHO scale).

Secondary objectives:

Evaluate limiting adverse events free survival (EIL) "severe" and "late", related to treatment.; to evaluate the disease-free survival of the treated site; to evaluate the intracranial disease-free survival (absence of new metastases); to evaluate the antitumor efficacy assessed by morphological objective response (complete response and partial response) to treatment by RECIST.

The objective of this study is to demonstrate the ability to deliver reliable, secure and efficient radiation by synchrotron radiation under dosimetry conditions similar to the techniques of advanced radiation therapy with high-energy photons. It will thus be a "platform" for future experimental test of new concepts of combined treatment with in situ administration of vectors molecules of heavy atoms by CED.

This is a study without any control group that will evaluate each patient's response according to RECIST criteria and record limiting adverse events (EIL), acute and late, by an independent external evaluation. Patients will have an initial phase of radiation at the ESRF to be followed by an additional irradiation at the University Hospital.

The study will be carried out in several successive steps, each including the number of patients needed to achieve the proposed objective. The number of patients will be three for each increment, unless extended for a particular level because of toxicity. Assuming an uneventful progression of the entire protocol described below, a total of 50 patients are to be included in this study in two to three years.

These steps are:

* Verification of the reproducibility of the kinetics of iodinated contrast in the tumor.
* Introduction of an iodinated contrast agent IV with a single-dose irradiation by SR.
* Dose escalation (Iodine and SR) and fractionation.
* Introduction of a platinum-injection system with the ultimate optimized RS protocol.
* Optimizing the dose of platinum by an advanced method of administration (CED or double platinum protocol).

The transition from one step to the next will be dependent on the feasibility of the previous step, the frequency and severity of side effects occurred at each step of the protocol. An External Review Committee will monitor the progress of the study and propose appropriate changes or discontinuation of the trial if appropriate.

The ESRF and the CHU of Grenoble have settled a cooperation agreement since the building of ESRF in the 80ties to develop medical application of SR: "RSRM". In 2003 the scientific team of the CHU and the University Joseph Fourier of Grenoble become an INSERM unit devoted to RSRM with the experimental medical imaging and radiotherapy with SR as a main goal: the different research axis of the Unit have been organized to contribute to these two domains and for each a specific department of the CHU has been associated. For the experimental medical imaging: the neuro-radiology and the cardiology departments; for experimental radiotherapy: the radiation oncology department of the CHU. That one is tidily associated: the patients will be selected, recruited, hospitalized, imaged and treated under the responsibility of the MD and the medical physicists of this CHU department and the patients will be transported for irradiation at the experimental irradiation room at ESRF for a part of their irradiation plan. This way, this first attempt of SR application to cancer treatment is completely embedded in the scientific and technical development of SR at ESRF which has invested large amount of money since years to modify, upgrade and equipped its biomedical facility.

This pioneer activity is followed by an industrial development of know how to make possible the future use of SR if it should issue significant and valuable progress. This effort, so far, has given way to the ThomX project.

ELIGIBILITY:
Inclusion Criteria:

* Controlled tumor disease in the primary site and no syndrome metastatic extracranial threatening short-term
* Presence of 1 to 3 metastases brain symptomatic or not, metachronous primary cancer of a solid, proven itself by histopathological examination
* In case of multiple lesions sites must be sufficiently spaced so that the PTV can be in separate horizontal planes
* PS < 2

Exclusion Criteria:

* One or more lesions > 3 cm in diameter on MRI, or infratentorial location
* Performed surgical resection or formal indication
* In progress or finished chemotherapy within the last 4 weeks
* Partial or total irradiation of brain in the past , or total body irradiation
* Presence of a second cancer that would be likely to render uncertain the identification of the origin of metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Safety | 5 years
  number of participant with adverse event (grade greater than 2), each adverse event will be gradueted according to Common Terminology Criteria for Adverse Events (CTCAE)Version 4.0

SECONDARY OUTCOMES:
Survival without limiting adverse events | 5 years
  Evaluate survival without limiting adverse events (EIL) "severe" and "late", related to treatment with score SOMA-LENT (grade greater than 2).
Acceptability | 2 years
  percentage of treated patients compared to the number of patients included
Treatment efficacy | 5 years
  Patients may be enrolled on study with measurable disease based on the RECIST, version 1.1. Disease assessment will be undertaken at baseline and then every month after treatment by MRI. Patients will be evaluated for response according to RECIST, v 1.1 guidelines.
  (Eisenhauer et al. 2009).
Quality of life | 5 years
  assessment with questionnary QLQ C30 and QLQ BN20 of EORTC

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Balosso, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Esrf / Id17, Grenoble, France

REFERENCES:
- See also: University Hospital of Grenoble — http://www.chu-grenoble.fr/